CLINICAL TRIAL: NCT01497288
Title: An Open Label, Randomised, Single-centre, Two Sequence, Cross-over Trial to Investigate the Pharmacokinetics (PK) of Single Doses of 200 µg, 400 µg and 2 x 400 µg of Intranasal Fentanyl Spray (INFS) in Healthy Subjects Using a Population PK Approach
Brief Title: A Trial to Investigate the Pharmacokinetics (PK) of Single Doses of 200 µg, 400 µg and 2 x 400 µg of Intranasal Fentanyl Spray (INFS) in Healthy Subjects
Acronym: PK400 INFS
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Takeda (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: FT-1301-101-RD; 2011-002549-37 (EudraCT Number); U1111-1135-2623 (Registry Identifier: WHO)
Record Dates: First submitted 2011-12-08; First posted 2011-12-22 (Estimated); Last update posted 2012-10-02 (Estimated); Status verified 2012-09

CONDITIONS: Healthy Volunteers
Keywords: Intranasal fentanyl spray; Population PK

ARMS (2):
- Sequence 1 (A-B-C) (Experimental): * A: single dose of 200 μg INFS (100 μL) (Instanyl®), administered on Day 1
  * B: single dose of 400 μg INFS (100 μL), administered 4 hours after the first treatment
  * C: two single doses of 400 μg INFS (100 μL) (10 min apart), administered 24 hours after the first treatment (Day 2)
  Interventions: Drug: INFS (Intranasal Fentanyl Spray)
- Sequence 2 (A-C-B) (Experimental): * A: single dose of 200 μg INFS (100 μL) (Instanyl®), administered on Day 1
  * C: two single doses of 400 μg INFS (100 μL) (10 min apart), administered 4 hours after the first treatment
  * B: single dose of 400 μg INFS (100 μL), administered 24 hours after the first treatment (Day 2)
  Interventions: Drug: INFS (Intranasal Fentanyl Spray)

INTERVENTIONS:
Drug: INFS (Intranasal Fentanyl Spray) — Intranasal Fentanyl Spray
  Other Names: (Instanyl®)

SUMMARY:
The overall clinical trial objective is to gain information about the Pharmacokinetics (PK) of a 400 µg dose strength of INFS using a Population PK (PopPK). In total, 20 healthy male and female subjects are planned to be randomized in the trial. Subjects will be randomized to one of two treatment sequences and treated with 3 different dosages (either 200 µg/dose INFS, 400 µg/dose or 400 µg two doses administered 10 minutes apart) over two days. Subjects will be hospitalized over a period of total 5 days, where safety assessments and pharmacokinetic samplings will be conducted.

ELIGIBILITY:
Eligibility Criteria:

Healthy male and female Caucasian or Black subjects between 18 and 55 years with a body mass index of 18-28 kg/m2 and a minimum weight of 50 kg.

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 20 (Estimated)
Dates: Start 2011-11; Primary Completion 2011-12 (Actual); Study Completion 2011-12 (Actual)

PRIMARY OUTCOMES:
Area Under the Curve From Time Zero to Extrapolated Infinite Time [AUC (0 - inf)] | Blood sampling for PK will be performed until 72 hours after the first treatment administration
  AUC= Area under the plasma concentration versus time curve (AUC) from time zero (pre-dose) to extrapolated infinite time (0 - inf). It is obtained from simulated single dose concentration time profiles derived from the final parameters of the PopPK model [clearance (CL), absorption rate constant (KA), central volume (V2), and bioavailability (F1)].

CONTACTS AND LOCATIONS:
Locations (1):
- Nycomed Investigational Site, Mannheim, Germany